CLINICAL TRIAL: NCT02190877
Title: A Study for Monitoring Subjects With Fluid-Management Issues Using Repeated Measurements In the Home Environment
Brief Title: Monitoring Subjects With Fluid-Management Issues In the Home Environment
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Perm-IRB-001
Record Dates: First submitted 2014-07-10; First posted 2014-07-15 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Heart Failure; Hypertension
Keywords: Heart Failure; Impedance; Fluids
MeSH Terms: conditions — Heart Failure; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Subjects taking diuretic medication: All subjects will be in the same group, Cohort 1

SUMMARY:
This study is designed to validate ease-of-use for the CoVa Monitoring System, along with simple statistical parameters such as reproducibility and inter-subject agreement between test and reference devices.

DETAILED DESCRIPTION:
The study has the following objectives:

Objective 1: investigate ease-of-use associated with the CoVa Monitoring System: determine if subjects could use the test device on a daily basis, and if the components of this system (Sensor, Gateway, Web-based System) were indeed operational

Objective 2: determine if daily application of the Sensor's adhesive Electrodes resulted in any skin irritation

Objective 3: determine that the long-term reproducibility of measurements made by the test device is as good or better than the long-term reproducibility of the reference device

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 21 (twenty-one) and 90 (ninety) years of age at screening.
* Subject will have a current prescription for a diuretic medication.
* Subject and/or legally authorized person/representative is willing to undergo the Informed Consent process prior to enrollment in the study.
* Subject is a candidate for this study based on the PI's opinion and knowledge of the subject's condition.

Exclusion Criteria:

* Subject is participating in another clinical study that may affect the results of either study.
* Subject is unable or not willing to wear electrode patches as required.
* Subject has skin sensitivity to adhesive or hydrogel materials used in electrode patches.
* Subject has a pacemaker, implanted cardioverter-defibrillator, or ventricular assist device.
* Subject is considered by the PI to be medically unsuitable for study participation.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be volunteers from Riverside Meadows Estates. Subjects will be taking one or more diuretic medication(s) prescribed by a physician
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Ease of Use | Each subject will be measured once per weekday over a 6 week period
  Investigate ease of use associated with the CoVa Monitoring System: determine if subjects could use the test device on a daily basis, and if the components of this system (Sensor, Gateway, Web-based System) were indeed operational

SECONDARY OUTCOMES:
SKin irritation and reproducibility | Each subject will be measured once per weekday over a 6 week period
  Determine if subjects had skin irritation from daily use for 30 days. Determine the long-term reproducibility of the measurements from the test device versus the reference device

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Banet, PhD, Principal Investigator — Baxter Healthcare Corporation
Locations (1):
- Riverside Meadows, Riverside, California, United States